CLINICAL TRIAL: NCT03780413
Title: Randomized Controlled Trial of PR-ESSENCE - an Intervention Model for Young People With Explosive and Challenging Behavior
Brief Title: PR-ESSENCE for Youth With Challenging Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Mats Johnson, MD PhD, Göteborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GNC PR-ESSENCE
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Behavior Problem of Childhood and Adolescence

STUDY DESIGN:
Intervention Model Description: RCT in which participants are randomized to active group (PR-ESSENCE for 10 weeks) or control group (treatment as usual for 10 weeks, followed PR-ESSENCE for 10 weeks)
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR-ESSENCE treatment (Active Comparator): The treatment group receives PR-ESSENCE for 10 weeks. Outcome measures are collected pre- and post-treatment, and after 6 months and one year.
  Interventions: Behavioral: PR-ESSENCE treatment
- Control (TAU) (Active Comparator): The control group receives 10 weeks of "treatment as usual (TAU)" (that is the standard psychoeducation, support and treatment given to all youth after neuropsychiatric assessment at our clinic), followed by 10 weeks of PR-ESSENCE. Outcome measures were collected pre- and post-treatment, and after 6 months and one year.
  Interventions: Behavioral: Control (TAU)

INTERVENTIONS:
Behavioral: PR-ESSENCE treatment
  Arms: PR-ESSENCE treatment
Behavioral: Control (TAU)
  Arms: Control (TAU)

SUMMARY:
The method "Collaborative and Proactive Solutions" (CPS) was developed by Dr. Ross Greene, Harvard University, to understand and help kids with social, emotional, and behavioral challenges. The underlying theory is that challenging behavior is caused by lagging cognitive skills, commonly in the domains of flexibility/adaptability, frustration tolerance, and problem-solving. Thus, challenging behavior can be seen as a form of developmental delay, and the most effective way for adults to help the children and to facilitate interaction with them is to understand the lagging skills behind the behavior and to change their own mindset accordingly.

ADHD and autism belong in a group of overlapping neurodevelopmental conditions now often referred to under the umbrella term of ESSENCE (Early Symptomatic Syndromes Eliciting Neurodevelopmental Clinical Examinations). A common impairing problem in both autism and ADHD - and in several of the other disorders in the group of ESSENCE (including Tourette syndrome and other tic disorders) - is the marked inability to control temper, coupled with oppositional-defiant behaviors.

The CPS-method has been evaluated by Ross Greene et al. in United States studies for families, in schools, and in institutions for young people with serious behavior problems. Our research group published the first Swedish study with the method in 2012, a small open pilot study. Based on experiences in clinical work after that study our group reached the conclusion that, in order for the intervention to be useful for families with severely impairing ESSENCE, the CPS model needed to be modified. After a number of research meetings and seminars, we therefore designed a new model, based on our CPS-experience, that we now refer to as PR-ESSENCE (Problem Resolution in ESSENCE).

The present study is a randomized controlled trial for approximately 130 children and adolescents aged 5-18 years, with neuropsychiatric disorders (for instance Attention Deficit Hyperactivity Disorder (ADHD), Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), Autism Spectrum Disorder (ASD), Tourette syndrome, learning difficulties), children who have been assessed at our Child Neuropsychiatry Clinic (CNC), and from the Habilitation Services, Child Psychiatry Units or schools in the Göteborg region.

DETAILED DESCRIPTION:
The "Collaborative Problem Solving" model was developed by Greene for the treatment of youth with oppositional behavior, and is now called Collaborative & Proactive Solutions (CPS). The aim of CPS is to help caregivers and children practice and learn problem solving strategies in collaboration. The theoretical base of the model is that problematic behavior is mainly caused by lagging skills, especially regarding frustration tolerance, flexibility and problem solving ability. The CPS model engages both the child and the parents in training, and may therefore have potential to give long-term improvement of lagging skills in handling problematic situations and to change the mindset towards strategies of mutual problem solving.

The CPS model was evaluated in a United States trial comparing CPS to Barkley's Parent Management Training program (PMT) in 47 children aged 4-12 years with ODD and affective dysregulation. Outcomes were similar between the two methods in most measures post-treatment and at 4 months follow-up. A recent larger randomized controlled US trial enrolled 134 children with ODD, aged 7 - 14 years, who were randomized to three groups (CPS, PMT or Waitlist Control). Both treatment groups had equivalent results in treatment response and remission of diagnostic status (50% were much to very much improved and no longer met diagnostic criteria), and both were superior to the WLC condition.

The first Swedish study of CPS, published by our research team 2012, was a small open pilot trial of 3 months CPS for 17 families and children aged 7-13 years, with ADHD, ODD and explosive behavior, showed promising results. At post-treatment 53% of the children were much or very much improved on global symptom and function ratings (Clinical Global Impression-Improvement; CGI-I rating 1-2), and after another 6 months when the children with severe residual ADHD symptoms also had received stimulant medication, 81% reached CGI-I levels of 1-2.

Thus previous research has suggested that CPS is an effective treatment for ODD in youth, but effectiveness in samples of children with various neurodevelopmental disorders has not yet been documented. Oppositional and explosive behavior is a major problem among youth with neurodevelopmental disorders and the demand for treatment strategies is great.

Experiences from treatment of children with complex neurodevelopmental disorders - ESSENCE (mainly including autism) have led the therapists in our team to make ESSENCE-adapted modifications to the CPS model, particularly regarding communication, structure, predictability, and focusing on the child's interests to facilitate interaction. We therefore designed a new model, based on our CPS-experience, that we now refer to as PR-ESSENCE (Problem Resolution in ESSENCE). During the early phases of this study, Dr. Greene gave advice and supervision to our treatment team, and the whole PR-ESSENCE model would not have been developed without this input.

Research questions

1. Can the PR-ESSENCE model reduce problematic behaviors? Outcome measures are the rating scales Swanson, Nolan and Pelham scale (SNAP-IV), Family Burden of Illness Module (FBIM), Eyberg Child Behavior Inventory (ECBI), Clinical Global Impression-Severity scale (CGI-S), Clinical Global Impression-Improvement scale (CGI-I) (see below).
2. Can the PR-ESSENCE model contribute to solve specific problem situations. Outcome measure is a Problem Rating Scale developed for this study
3. Can the PR-ESSENCE model improve psychiatric well-being and self-image in the participants? Outcome measure is the Beck Youth Inventories.

Method The present study is designed to investigate how well PR-ESSENCE works for challenging behaviors in well-defined clinical samples of children with complex neurodevelopmental disorders. Participants are children and adolescents aged 5-18 years, with any neurodevelopmental diagnosis, and with intellectual level in the normal range.

After neuropsychiatric assessment and diagnosis at our centre or at the Child Psychiatry Centres in Gothenburg 130 children and adolescents aged 5-18 years with complex neurodevelopmental disorders (i.e. autism, ADHD, learning disorders, dyslexia, tics, and Conduct Disorder) and problematic behaviors are invited to participate in the trial. They are randomized to a PR-ESSENCE treatment group and a control group. The treatment group receives PR-ESSENCE for 10 weeks. The control group receives 10 weeks of "treatment as usual (TAU)" (that is the standard psychoeducation, support and treatment given to all youth after neuropsychiatric assessment at our clinic), followed by 10 weeks of PR-ESSENCE. Outcome measures are collected pre- and post-treatment, and after 6 months and one year. During the PR-ESSENCE treatment period the parents and children meet the therapists at approximately 10 visits, at which they collaborate to find problem solving strategies, which they then practice at home between visits.

Inclusion criteria

1. Children and adolescents aged 5-18 years with neurodevelopmental disorders and serious problematic behaviors.
2. Intellectual function in the normal range, according to WISC-test and clinical judgment
3. Participants taking psychoactive medication can be included if the medication has been unchanged for at least one month before baseline, and remains unchanged during the treatment period.

Exclusion criteria

1. Bipolar disorder, psychosis, or other unstable psychiatric or medical disorder which in the investigator's judgment makes participation in the trial unsuitable.
2. Substance use.

Outcome measures The following measures are collected at baseline (pre-treatment), after the treatment/TAU period (post-treatment), after 6 months (6-month follow-up) and 1 year (one-year follow-up). To obtain results from different perspectives ratings from four sources were used, i.e. ratings by independent blinded assessors, and by parents, children and therapists.

Rating of independent blinded assessor CGI-I: Scale for global rating of improvement or deterioration of problems/symptoms (scale from 1-7; 1 very much improved, 7 very much worse) CGI-S: Scale for global rating of problem/symptom severity (scale from 1-7; 1 no problems, 7 very severe problems)

Parent ratings SNAP-IV - rating scale for ADHD symptoms FBIM - rating scale of family stress/burden ECBI - rating of behavior problems

Child self-rating Beck Youth Inventories: For rating of depression, anxiety, irritability, externalizing behavior, and self image (child interviewed).

Therapist ratings Problem Rating Scale (in which the severity of the problematic situations before and after treatment is rated)

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents aged 5 to18 years with neuropsychiatric diagnoses and serious challenging behaviors/explosive reactions.
2. Intellectual function in the normal range, according to WISC-test, adaptive function and clinical judgment.
3. Participants treated with psychoactive medication (e.g. for ADHD) can be included if the medication has been unchanged during at least one month prior to baseline, and is unchanged during the treatment period.

Exclusion Criteria:

1. Bipolar disorder, psychosis, or other unstable psychiatric or medical condition that according to the investigators opinion makes study participation unsuitable.
2. Substance Use.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
CGI-S/CGI-I change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Clinical Global Impression - Severity and Improvement (by blinded assessor). Range 1-7 points, lower is better. A global assessment of severity and change in behavior problems and everyday function.

SECONDARY OUTCOMES:
ODD Scale change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Oppositional Defiant Rating Scale (Ross Greene's), parent-rated. An assessment of DSM-5 Oppositional Defiant Disorder symptoms. Range 34-170, lower is better.
SNAP-IV change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Rating scale of ADHD symptoms (parent-rated). Range 0-54 Points, lower is better.
FBIM change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Family Burden of Illness Module (measure of family stress - parent-rated). Range 0-24, lower is better.
ECBI change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Eyberg Child Behavior Inventory (measure of behavior problems, parent-rated). Range 0-216, lower is better.
RPQ change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Relationship Problems Questionnaire (measure of relation and attachment, parent-rated). Range 0-30 Points, lower is better.
Beck's Youth Inventory change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Self-rating of depression, anxiety, irritability, behavior problems, and self-image. Self-rated by interview. Range 0-300, lower is better.
Problem solving scale change | Baseline, post-treatment/control period (3 months), 6 months and 1 year post-treatment
  Measures number and type of problem situations solved (therapist-rated). Range 0-infinite number, higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gillberg, Professor, Study Chair — Gillberg Neuropsychiatry Centre, Goteborg University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson M, Gillberg C, Vinsa I, Fransson G, Samuelsson L, Jakobsson K, Ostlund S, Fernell E, Gillberg C. A randomized controlled trial of a new intervention in early symptomatic syndromes eliciting neurodevelopmental clinical examinations: PR-ESSENCE. Eur Child Adolesc Psychiatry. 2023 Jan;32(1):63-74. doi: 10.1007/s00787-021-01837-z. Epub 2021 Jul 3. PMID 34218336